CLINICAL TRIAL: NCT00876538
Title: A Double Blind, Placebo Controlled Study of the Effect of 330 mg QD of TRO19622 in the Treatment of Chemotherapy Induced Peripheral Neuropathy
Brief Title: Effect of TRO19622 in the Treatment of Patients With Chemotherapy Induced Peripheral Neuropathy
Acronym: CIPN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WN29851; EudraCT number: 2008-001218-26; TRO19622 CL E Q 1204-1 (Other: trophos id)
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy
Keywords: Chemotherapy Induced Peripheral Neuropathy; TR019622; Trophos
MeSH Terms: interventions — olesoxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRO19622 (Experimental): 2 capsules of TRO19622 (330mg) once day with the noon meal
  Interventions: Drug: Olesoxime (TRO19622)
- Control (Placebo Comparator): 2 capsules of placebo once day with the noon meal
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Olesoxime (TRO19622) — 2 capsules of TRO19622 (330 mg) once day with the noon meal
  Arms: TRO19622
Drug: Placebo Control — Placebo Control 2 capsules once day with the noon meal
  Arms: Control

SUMMARY:
The purpose of this study is to test the effect of TRO19622 on peripheral neuropathy scores after 6 weeks treatment and is based on the separate assessment of pain and dysesthesia scores.

DETAILED DESCRIPTION:
Chemotherapy Induced Peripheral Neuropathy represents a frequent and invalidating side effect that requires treatment. Current treatment options are multiple, but none have yet demonstrated efficacy in double-blind clinical trials .

This study will provide information useful to determine the potential of TRO19622 to relieve both pain and dysesthesia which are the most common symptoms experienced by patients with peripheral neuropathy following taxane chemotherapy.

At the start of the study, patients will be randomized to one of two groups : TRO19622 (330 mg QD or placebo once a day).

Each treatment will be administered for 6 weeks. Additionally, patients will have the option to continue treatment for another 6 weeks duration.

Treatment will be administered under double-blind conditions. The product under evaluation will be administered to patients receiving the standard of care for CIPN.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an Informed Consent to participate to the trial before any study related procedure has taken place.
* Be >18 years and if a female with adequate contraception if of child bearing potential.
* Have paclitaxel (or other taxane) induced peripheral neuropathy assessed by the presence of a NCI-CTC version 2 neuropathy sensory grade >/= 2 .
* Peripheral neuropathy as clinically diagnosed during the neurological examination including sensitivity, motor function and deep tendon reflex assessments
* With Neuropathic pain as assessed by the presence of measurable pain perception (previous 24h)on the Likert numerical rating scale >/= 4 points at the screening visit and confirmed on DN4 with a score >/= 4 and/or Dysesthesia as assessed by the presence of measurable dysesthesia (previous 24h) on the Likert numerical rating scale >/= 4 points at the screening visit
* Persistent neuropathy for at least 3, but no more than 12 months after the end of chemotherapy.
* Be either pain treatment naive or have important side effects or inadequate relief from their current pain medication (stable over last month).

The following inclusion criteria should be ascertained at the baseline visit:

* Peripheral neuropathy symptoms: Have measurable pain perception (previous 24h) on the Likert numerical rating scale with a mean >/= 4 points calculated from at least 4 daily measurements over the 7 days immediately prior to the Baseline Visit and/or Dysesthesia as assessed by the presence of measurable dysesthesia with a mean >/= 4 points calculated from at least 4 daily measurements over the 7 days immediately prior to the Baseline Visit.
* Have an electrocardiogram (ECG) at Baseline without any clinically significant abnormality.
* Have an expected survival > 6 months.

Exclusion Criteria:

* Have a documented neuropathy or risk factors of neuropathy which might interfere with the assessment of the severity of pain (eg, including, but not limited to, type 2 diabetes, peripheral vascular disease, B12 Vitamin deficiency, thyroid dysfunction, post surgical neuropathic pain, post-traumatic neuropathy, or neuropathy in relation with disease progression).
* Have other neurological diseases that may produce weakness, sensory loss, or autonomic symptoms, or laboratory test abnormality.
* Refractory to treatment defined as not improved, according to the Investigator, by 3 or more treatments prescribed for the current PN symptoms.
* HIV positive serology.
* History of, or current cardiac dysrhythmias and / or a history of cardiovascular disease,including myocardial infarction, except patients with only well controlled hypertension.
* Have had prior (within the past 6 months) or have concurrent neurotoxic drugs (e.g., but not limited to, cisplatin, vincristine, vinblastine, cytarabine, thalidomide, bortezomib, or procarbazine, capecitabine, navelbine).
* Have a current medication that may have a similar mechanism of action as TRO19622: acetyl-L-carnitine
* Have a current medication that could interfere with TRO19622 pharmacokinetics: tamoxifen
* Have current medications that could interfere with TRO19622 absorption such as ezetimibe, bile salts chelators, fibrates, phytosterols, fish oils.
* Have a current medication of lipid lowering agents other than statins.
* Have a recent history (within the previous 6 months) or current evidence of alcohol or drug abuse.
* Have concurrent unstable disease involving any system (eg, advanced carcinoma other than carcinoma justifying the recent treatment with taxanes, myocardial infarction, clinical or ECG signs of myocardial ischemia, cardiac insufficiency, anginal symptoms, current symptoms of CAD, renal impairment, or any other condition that in the opinion of the Investigator would make the patient unsuitable for study participation)
* Be pregnant female or lactating.
* Have renal impairment defined as blood creatinine > 1.5× upper limit of normal (ULN)
* Hemostasis disorders or current treatment with oral anticoagulants.
* Have hepatic impairment hepatic function as follows: liver enzymes (ALT and AST) > 2× ULN or > 3.5× ULN in case of liver metastasis
* Are not able to comply with regard to the known contraindications, warnings and precautions, drug-interactions and dosing recommendations of paracetamol or tramadol.
* Be possibly dependent on the Investigator or the Sponsor (eg, including, but not limited to, affiliated employee).
* Participated in any other investigational drug or therapy study with a non approved medication,within the previous 3 months.
* Known hypersensitivity to one of the capsules' ingredients
* Any other condition which, in the opinion of the investigator would impede competence or compliance or possibly hinder completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the measure of the percentage of responders defined as patients with a minimum decrease of 50 % of their maximum neuropathic pain dimension (either pain or dysesthesia) present at baseline. | The mean pain score during the last 7 days of the treatment period will be compared to the mean score of the last 7 days of the screening score period.

SECONDARY OUTCOMES:
Assessment with respect to placebo of the effect of TRO19622 on Neuropathic Pain Inventory Score(total and by dimension) | Screening visit; V0; V1; V2; V3; V4 ; V5
Assessment with respect to placebo of the effect of TRO19622 on Short- Form BPI | Screening visit; V0; V1; V2; V3; V4 ; V5
Assessment with respect to placebo of the effect of TRO19622 on Quality of life questionnaire (CIPN 20) | V0; V3; V5
Assessment with respect to placebo of the effect of TRO19622 on Dysgueusia questionnaire | V0; V3; V5
Assessment with respect to placebo of the effect of TRO19622 on Quantitative Sensory Testing | V0; V3; V5
Assessment with respect to placebo of the effect of TRO19622 on ENMG | V0; V3; V5
Assessment with respect to placebo of the effect of TRO19622 on the use of rescue medication | Screening visit; V0; V1; V2; V3; V4 ; V5
Assessment with respect to placebo of the effect of TRO19622 on safety profile | Screening visit; V0; V1; V2; V3; V4 ; V5
Assessment with respect to placebo of the effect of TRO19622 on Global Impression of change as assessed by Investigator | V1; V2; V3; V4; V5
Assessment with respect to placebo of the effect of TRO19622 on Global Impression of change as assessed by patient | V1; V2; V3; V4; V5
Assessment with respect to placebo of the effect of TRO19622 on Hospital Anxiety and Depression scale | V0;V3;V5

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Krakowski, MD, Principal Investigator — Centre Alexis Vautrin / Département d'Oncologie Médicale/ Nancy
Locations (8):
- France (8):
  - Centre Hospitalier de Versailles Hôpital André Mignot Service d'Hématologie-Oncologie, Le Chesnay
  - Centre Oscar Lambret Département de Sénologie, Lille
  - Centre Léon Bérard Département de Soins de Support, Lyon
  - C.R.L.C Val d'Aurelle Service d'Oncologie Médicale, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Centre Antoine Lacassagne, Nice
  - Hôpital Nord CHU Saint Etienne Centre de la douleur, Saint-Etienne
  - Hôpital Privé de l'Ouest Parisien Service d'Oncologie, Trappes